CLINICAL TRIAL: NCT05086432
Title: Sputum Cytometry Guided Management for the Elimination of Chronic Cough in Patients With Interstitial Lung Disease (SpECC-ILD) - a Randomized Controlled Trial
Brief Title: Sputum Cytometry Guided Management for the Elimination of Chronic Cough in Patients With ILD
Acronym: SpECC-ILD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); Vitalograph (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13513
Record Dates: First submitted 2021-09-28; First posted 2021-10-20 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2024-11

CONDITIONS: ILD
Keywords: ILD; Sputum; Chronic cough
MeSH Terms: conditions — Chronic Cough | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sputum-guided management (Experimental): During Weeks 0 to 16, participants randomized to the intervention arm will receive open-label sputum-guided management of airway inflammation (Table 1 in protocol) identified during screening (Figure 2 in protocol). Airway eosinophilia will be treated with regular inhaled corticosteroids based on the severity of eosinophilic inflammation. In participants with airway neutrophilia, as per the standard of care, sputum culture and sensitivity will be sent, and pathogenic organisms treated. Those participants with airway neutrophilia with negative cultures will be treated with thrice weekly Azithromycin (250mg). Combined eosinophilia and neutrophilia will receive treatment with both ICS and Azithromycin as per Table 2 in protocol.
  Interventions: Other: Sputum-guided management
- Standard of Care (Active Comparator): Participants in this arm will receive standard of care treatment as determined by their ILD specialist who will be blinded to the results of the sputum analysis.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Sputum-guided management — As previously described.
  Arms: Sputum-guided management
Other: Standard of Care — As previously described.
  Arms: Standard of Care

SUMMARY:
In Interstitial Lung Disease (ILD) there is thickening of lung tissue, which makes it difficult for patients to breathe and get enough oxygen into their bodies. In addition to shortness of breath, daily cough is very common, with 4 out of 5 patients experiencing this symptom. Cough in particular has a major impact on the ability to exercise, be active, and to simply enjoy life.

There are many reasons for cough in ILD, and very often there are multiple overlapping causes. It is hard to improve cough in these patients, with available medicines providing limited relief. One explanation for this gap is an incomplete understanding of cough in ILD. To improve patients' cough there is a need to better understand its cause. In other lung diseases, such as asthma, doctors and scientists have used phlegm tests to measure inflammation in the lung, which helps them choose the right medicine for the right patient. This has not been done for ILD, even though it has recently been found that many patients with ILD and everyday cough have abnormal phlegm tests. Using this strategy in ILD could improve patients' cough and quality of life, and possibly even slow progression of the disease.

DETAILED DESCRIPTION:
SpECC-ILD is an open-label, randomized controlled trial assessing the efficacy of sputum-guided management (using sputum cytometry) compared to standard care over 16 weeks in patients with chronic cough and ILD.

A total of 80 participants will be enrolled and randomized in a 1:1 ratio to either sputum guided therapy or standard of care for a total of 16 weeks. Participants randomized to the intervention arm will receive open-label sputum-guided management of airway inflammation identified during screening. Participants in this arm will receive standard of care treatment as determined by their ILD specialist who will be blinded to the results of the sputum analysis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent consistent with ICH-GCP and local laws, signed prior to any study procedures being performed
* Age >18 years
* A clinical diagnosis of ILD with accepted specific diagnoses including:
* Idiopathic pulmonary fibrosis (IPF)
* Chronic hypersensitivity pneumonitis associated ILD (CHP-ILD)
* Connective tissue disease associated ILD (CTD-ILD)
* Pneumoconiosis
* Daily Cough for at least 8 weeks
* Able to produce an adequate sample with sputum induction

Exclusion Criteria:

* Patients with a diagnosis of systemic sclerosis associated ILD (SSc-ILD) or sarcoidosis
* Cause of cough attributed to a known etiology (ex. ACE-inhibitor, uncontrolled gastroesophageal reflux or upper airway cough syndrome, acute viral illness)
* Current use of inhaled corticosteroids
* Current use of systemic corticosteroids (prednisone equivalent > 20mg/day)
* Current use of chronic antibiotics
* Airflow obstruction (ie. pre-bronchodilator FEV1/FVC ratio < 0.7)
* History of physician-diagnosed asthma
* History of emphysema
* A history of cholestatic jaundice or hepatic dysfunction associated with prior use of azithromycin
* Moderate to severe hepatic dysfunction with a Child Pugh score >10
* Known allergy or hypersensitivity to inhaled corticosteroids or macrolide antibiotics
* Corrected QT-interval (QTc) on screening electrocardiogram (ECG) of > 450ms
* An established history of untreated atypical mycobacterial infection
* A history of hearing impairment, tinnitus, or vertigo
* Medication use likely to suppress cough (ex: morphine, gabapentin, amitriptyline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in hourly cough frequency | 16 weeks
  The difference in hourly cough frequency over a 24-hour period between baseline and end of study.

SECONDARY OUTCOMES:
Change in FEV1 | 16 weeks
  The difference in forced expiratory volume in 1 second (as obtained by spirometry) between baseline and end of study
Change in FVC | 16 weeks
  The difference in forced vital capacity (as obtained by spirometry) between baseline and end of study
Change in Leicester Cough Questionnaire | 16 weeks
  The difference in LCQ between baseline and end of study
Change in King's Brief ILD Questionnaire | 16 weeks
  The difference in KB-ILD between baseline and end of study
Change in sputum total cell count | 16 weeks
  The difference in sputum total cell count between baseline and end of study
Change in sputum neutrophils | 16 weeks
  The difference in sputum neutrophil percent between baseline and end of study
Change in sputum eosinophils | 16 weeks
  The difference in sputum eosinophil percent between baseline and end of study
Adverse events | 16 weeks
  Adverse events reported by participants
Serious adverse events | 16 weeks
  Serious adverse events reported by participants
Completion rates for Bi-weekly LCQ | 16 weeks
  Rates of completion for bi-weekly LCQ
Study medication adherence rate | 16 weeks
  Rates of adherence to study medications

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No